CLINICAL TRIAL: NCT00573027
Title: Coronary Microvascular Disease and Endothelial Function in Women and Men
Brief Title: Heart Disease of the Small Arteries in Women and Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 8221
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Heart Disease
Keywords: microvascular dysfunction; Microvascular
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): 1. fill out baseline demographic and health/medical history questionnaires, CV risk factors, reasons of diagnosis of ischemia, information of coronary artery, and medication use
  2. undergo clinically indicated coronary angiography with adenosine coronary flow reserve measurement and acetylcholine provocative testing in the cardiac catheterization laboratory (Appendix);
  3. undergo noninvasive Peripheral Artery Tonometry (PAT) testing (Appendix);
  4. undergo clinically indicated Cardiac Magnetic Resonance (CMR) imaging (Appendix) to detect subendocardial ischemia (if indicated and referred by the treating physician). The three tests (heart catheterization with adenosine coronary flow reserve testing, acetylcholine provocative vasomotor testing during heart catheterization, cardiac MRI) are performed for standard care.
  5. have blood and urine testing.
  6. fill out health questionnaires
  7. be followed prospectively 6-week, 6-month, and annually for clinical status
  Interventions: Procedure: noninvasive tests

INTERVENTIONS:
Procedure: noninvasive tests — clinically indicated coronary angiography with adenosine coronary flow reserve measurement and acetylcholine provocative testing in the cardiac catheterization laboratory; Peripheral Artery Tonometry (PAT) testing; Cardiac Magnetic Resonance (CMR) imaging.

SUMMARY:
Women suffer disproportionately than men from Cardiac Syndrome X ( chest pain in the absence of flow limiting coronary artery stenosis). Coronary microvascular disease is hypothesized to mediate chest pain in this syndrome. This disorder of the small heart vessels (arterioles) compared to the large vessels (arteries) is not diagnosed during routine heart catheterization. This results in delays in diagnosis, missed opportunities for treatment, and likely contributes to the increased death rate from coronary heart disease in women compared to men.

Current testing for small vessel disease is performed in the cardiac catheterization laboratory using specialized testing and is not performed routinely. Accordingly, women with this condition are either falsely reassured, or misdiagnosed as another non-cardiac condition. Unnecessary healthcare costs related to re-hospitalization and repeat angiography are incurred, while women are often not initiated on appropriate lifesaving treatment. We and others have demonstrated in randomized controlled trials that therapies that target the endothelium, e.g. statins, ACE inhibitors, and exercise are effective in this condition.

Majority of women with Cardiac Syndorme X go undiagnosed. Recent studies have shown significant increased health care costs, morbidity and mortality related to this disease. It is becoming more important to further characterize this group of patients and we hope to do that with our study.

DETAILED DESCRIPTION:
Study Aims:

1. To establish prevalence of microvascular disease in women and men with Cardiac Syndrome X
2. To study the predictive value and utility of noninvasive tests like Peripheral Artery Tonometry (PAT) and Cardiac Magnetic Resonance (CMR) in diagnosing Cardiac Syndrome X.
3. To establish prognosis in women and men with Cardiac Syndrome X.
4. To elucidate the risk factors, clinical features, diagnostic methods, treatment, and prognosis of patients with microvascular angina (MVA).

With this research study, we want to specifically study a group of patients who have chest pain or other signs or symptoms suggestive of heart disease but don't have visible blockages in the large heart arteries. Patients with chest pain who undergo heart catheterization but have no blockages of large heart arteries will be consented and enrolled. Patients will be asked to fill out questionnaires about their medical history, including family, reproductive and, social histories. They will also be asked to undergo testing during heart catheterization that would test for abnormalities in their small heart arteries using medications, acetylcholine and adenosine. This testing is a standard of care procedure given at the discretion of the treating physician. Patients would receive this test whether they participate in the research or not. The test is performed by infusing acetylcholine and adenosine through the same catheter that is used for routine heart catheterization. This test may add an additional 15 minutes to the heart catheterization procedure.

In addition, patients will be asked to undergo a non-invasive test called Peripheral Arterial Tonometry or PAT for research purposes and in some cases, if clinically indicated a Cardiac Magnetic Resonance (CMR) imaging test as a standard of care. Patients will be followed up using phone questionnaires at 6 months and than annually thereafter. It is proposed that problems with the function of the large and small arteries may be responsible for giving some patients their symptoms of chest pain and put them at risk for heart attacks. PAT may help us more easily and non-invasively measure this function by testing the arteries in the arm. Selected patients will also undergo CMR imaging that may be useful to detect abnormalities in the inner layer of the heart muscle resulting from the abnormal function of the large and small heart arteries. These non-invasive tests will be corroborated with results from invasive testing during heart catheterization, which is considered the gold standard for testing for function of the large and the small heart arteries.

The three tests (heart catheterization with adenosine coronary flow reserve testing, acetylcholine provocative vasomotor testing during heart catheterization, cardiac MRI) are performed for standard care.

Blood and urine collection have been added to this protocol as a secondary outcome for future tests and for testing whether impaired Endothelial Progenitor Cell (EPC) number is related to the presence and severity of microvascular disease.

Results from our study will help confirm the need to test patients with chest pain and open large arteries during heart catheterizations for abnormalities in the function of the large and small heart arteries, and to validate the usefulness of using non-invasive techniques like PAT and CMR for detecting this problem. The study will also help confirm the increased risk of heart attack associated with the abnormal function in the large and small arteries in these patients.

Subjects will be asked if they are interested in receiving information on Pro00015124 (repository/collection). If they are interested, they will be consented under Pro00015124. No specimens collected as part of this study will be forwarded to Pro00015124.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men with signs and symptoms of myocardial ischemia and angina or angina equivalent (chest pain, abnormal stress testing, abnormal noninvasive testing) or microvascular angina (MVA) which is defined as angina and ischemic ECG changes without organic obstructive stenosis or epicardial spasm of the coronary arteries
2. No obstructive coronary artery disease performed within the previous 24 months (<50% luminal obstruction in one or more coronary arteries on angiography).
3. Age > 18 years old
4. Competent to give informed consent

Exclusion Criteria:

1. Obstructive CAD ≥ 50% luminal diameter stenosis in ≥ 1 epicardial coronary artery,
2. Acute coronary syndrome (defined by the ACC/AHA criteria, Braunwald 2000),
3. Primary valvular heart disease clearly indicating the need for valve repair or replacement;
4. Patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support;
5. Prior or planned percutaneous coronary intervention or CABG or prior acute MI in prior 30 days;
6. Prior non-cardiac illness with an estimated life expectancy <4 years;
7. Unable to give informed consent;
8. Chest pain with a non-ischemic etiology (e.g.,pericarditis, pneumonia, esophageal spasm);
9. Contraindications to adenosine or Regadenoson (Lexiscan)
10. Women and men with intermediate coronary stenoses (>20% but <50% luminal diameter stenosis assessed visually at the time of angiography) will undergo clinically indicated IVUS testing based on the judgment of the operator; those determined to have flow FFR or obstructing stenosis will be excluded from the overall study.
11. Heart failure (NYHA Class III or IV on treatment)
12. LV dysfunction (ejection fraction <40%)
13. Documented obstructive myocardiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2005-11; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
noninvasive Peripheral Artery Tonometry (PAT) testing and Cardiac Magnetic Resonance (CMR) imaging for the outcome of coronary endothelial dysfunction | 120 minutes

SECONDARY OUTCOMES:
clinically indicated coronary angiography with adenosine coronary flow reserve measurement and acetylcholine provocative testing | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: C.Noel Bairey-Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No